CLINICAL TRIAL: NCT04607512
Title: A Three-Way Crossover Study to Evaluate the ECG Effects of Telaglenastat in Healthy Adult Subjects
Brief Title: Study to Evaluate the ECG Effects of Telaglenastat in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CX-839-013
Record Dates: First submitted 2020-10-20; First posted 2020-10-29 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Cardiac Safety

STUDY DESIGN:
Intervention Model Description: double-blind (with respect to telaglenastat and placebo), placebo- and positive controlled, 3 way crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: telaglenastat, placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Telaglenastat (Experimental): 800 mg telaglenastat (4 x 200 mg tablets) administered twice daily (BID) on Days 1 3, with a single dose administered on the morning of Day 4
  Interventions: Drug: telaglenastat
- Telaglenastat Placebo (Placebo Comparator): 800 mg placebo (4 x 200 mg tablets) administered twice daily (BID) on Days 1 3, with a single dose administered on the morning of Day 4
  Interventions: Other: telaglenastat placebo
- Moxifloxacin (Active Comparator): Single dose of 400 mg moxifloxacin (1 x 400 mg tablet) administered on the morning of Day 4
  Interventions: Other: moxifloxicin

INTERVENTIONS:
Drug: telaglenastat — glutaminase inhibitor
  Arms: Telaglenastat
Other: telaglenastat placebo — matching placebo for telaglenastat
  Arms: Telaglenastat Placebo
Other: moxifloxicin — positive control
  Arms: Moxifloxacin

SUMMARY:
This study is designed to evaluate the effects of telaglenastat on cardiac repolarization (relative to placebo) in healthy adult subjects.

DETAILED DESCRIPTION:
This is a multiple-dose, randomized, double-blind (with respect to telaglenastat and placebo), placebo- and positive controlled, 3 way crossover thorough QT (TQT) study in healthy adult subjects.

On Day 1 of Period 1, subjects will be randomized to 1 of 6 treatment sequences.

In Treatments A and B, subjects will receive the assigned treatment on Day 1 through the morning of Day 4. In Treatment C, subjects will receive a single-dose administration of moxifloxacin in the morning of Day 4. Cardiodynamic readings will be collected for 24 hours on Days 1 and 4. Plasma PK samples will be collected prior to dosing (for Treatments A and B or Hour 0 for Treatment C) and up to 24 hours on Days 1 and 4 of all treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female (of non childbearing potential only), 18-45 years of age, inclusive, at the screening visit.
2. Continuous non smoker who has not used nicotine containing products (chewed or smoked) or replacement products, including electronic cigarettes, for at least 3 months prior to the first dosing and throughout the study, and have a negative cotinine test result at the screening and check-in visits.
3. Body mass index (BMI) ≥ 18 and ≤ 28.0 kg/m2 at the screening visit.
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee.
5. A female of non childbearing potential has undergone one of the following sterilization procedures at least 6 months prior to the first dosing:

   * hysteroscopic sterilization;
   * bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy. or be postmenopausal with amenorrhea for at least 1 year prior to the first dosing and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status.
6. A non vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days after the last dosing. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to the first dosing. A male who has been vasectomized less than 4 months prior to study first dosing must follow the same restrictions as a non vasectomized male).
7. If male, must agree not to donate sperm from the first dosing until 90 days after the last dosing.
8. Able and willing to swallow whole tablets without breaking, cutting or chewing.
9. Understands the study procedures in the informed consent form (ICF) and is willing and able to comply with the protocol.

Exclusion Criteria:

1. History or presence of diseases which, as judged by the investigator, may affect the outcome of this study, including but not limited to significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, or neurologic disease.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of hospitalization for a major illness or procedure in the last 3 months. Subjects with preplanned and elective surgery or a procedure that requires inpatient hospitalization throughout the duration of the study are excluded from the study.
4. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or pose an additional risk to the subject by their participation in the study.
5. Any condition that may interfere with the absorption, metabolism, or elimination of telaglenastat.
6. Clinically significant laboratory values that would place the subject at undue risk in the opinion of the PI or designee, including but not limited to serum alanine aminotransferase (ALT) or serum aspartate aminotransferase (AST) > 1.2 × upper limit of normal at the screening visit.
7. History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing.
8. History or presence of hypersensitivity or idiosyncratic reaction to the study drug(s) or related compounds.
9. History of tendon disease/disorder related to quinolone treatment.
10. Female subjects with a positive pregnancy test at the screening visit or first check in or who are lactating.
11. Positive urine drug or alcohol results at the screening visit or first check in.
12. Regular use of alcohol within 6 months prior to the screening visit (more than 21 units of alcohol per week for men, or 14 units of alcohol per week for women [1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
13. Use of recreational drugs (such as marijuana) within three months prior to the screening visit or illicit drugs (such as cocaine or methamphetamine) within one year prior to the screening visit.
14. Positive results at the screening visit for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
15. Family history of QTc prolongation or of unexplainable sudden death at < 50 years of age.
16. History or presence of:

1. Risk factors for Torsade de Pointes (eg, heart failure, cardiomyopathy, or family history of Long QT Syndrome or Brugada Syndrome) 2. Sick sinus syndrome, second or third degree atrioventricular block, myocardial infarction, pulmonary congestion, symptomatic or significant cardiac arrhythmia, prolonged QTcF, or clinically significant conduction abnormalities 3. History of angina, myocardial ischemia, arrythmia, heart failure or stroke 4. Clinically significant cardiac history or presence of ECG findings as judged by the PI or designee at screening or first check in, including the presence of abnormal sinus rhythm (HR < 50 or > 100 bpm; measurement may be repeated once at the discretion of the PI or designee) 17. Resting supine blood pressure is less than 90/50 mmHg or greater than 140/90 mmHg at the screening visit (may be repeated twice at the discretion of the PI or designee).

18. Unable to refrain from or anticipates the use of:

* Any drug, including prescription and non prescription medications (including gastric acid reducing [PPIs, histamine-2 receptor antagonists] or buffering agents [eg Tums]), herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing and throughout the study. Medication listed as part of acceptable birth control methods will be allowed (refer to Section 11.1). After randomization/dosing, paracetamol (up to 2 g per 24 hours) may be administered at the discretion of the PI or designee.
* Any drugs known to be substrates of CYP2C9 (eg, warfarin) within 14 days prior to Day 1 and throughout the study. Appropriate sources (eg, Flockhart TableTM) will be consulted to confirm lack of PK/PD interaction with study drug.
* Food and beverages containing xanthines/caffeine (including energy drinks) for 24 hours prior to Day 1 of Period 1;
* Food and beverages containing alcohol for 48 hours prior to Day 1 of Period 1.
* Food and beverages containing grapefruit/Seville orange for 14 days prior to Day 1 of Period 1.

  19. Has been on a diet incompatible with the on study diet, in the opinion of the PI or designee, within the 30 days prior to the first dosing and throughout the study.

  20. Is lactose intolerant or has any significant food allergy, in the opinion of the PI or designee.

  21. Donation of blood or plasma, or significant blood loss within 90 days prior to the first dosing.

  22. Donation of bone marrow within the last 6 months prior to the first dosing. 23. Participation in another clinical study within 90 days prior to the first dosing. The 90 day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
To assess the effects of telaglenastat on cardiac repolarization (relative to placebo) using the therapeutic dose and schedule in healthy adult subjects | Plasma samples and triplicate ECGs taken on Days 1 and 4 of each period at baseline, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16 and 24 hours post administration
  Evaluation of the relationship between the plasma concentrations of telaglenastat and its metabolite 110826 with the ΔQTc, placebo-adjusted and corrected for HR based on the Fridericia QT correction method (ΔΔQTcF)

SECONDARY OUTCOMES:
To assess the effects of telaglenastat on heart rate (relative to placebo) using the therapeutic dose and schedule in healthy adult subjects. | Triplicate ECGs taken on Days 1 and 4 of each period at baseline, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16 and 24 hours post administration
  Time-point change from baseline in QTc, placebo-adjusted and corrected for HR based on the Fridericia QT correction method (ΔΔQTcF)
To assess the effects of telaglenastat on other ECG parameters (relative to placebo) using the therapeutic dose and schedule in healthy adult subjects. | Triplicate ECGs taken on Days 1 and 4 of each period at baseline, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16 and 24 hours post administration
  Placebo-corrected ΔHR, ΔQTcF, ΔPR, and ΔQRS (ΔΔHR, ∆∆QTcF, ΔΔPR, and ΔΔQRS) evaluated at each post baseline time point ('by time point' analysis)
To assess the effects of telaglenastat on changes of T-wave morphology and U wave presence (relative to placebo) using the therapeutic dose and schedule in healthy adult subjects. | Triplicate ECGs taken on Days 1 and 4 of each period at baseline, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16 and 24 hours post administration
  Frequency of treatment emergent changes of T-wave morphology and U wave presence
To demonstrate sensitivity of this QTc assay using moxifloxacin as a positive control. | Triplicate ECGs taken on Days 1 and 4 of each period at baseline, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16 and 24 hours post administration
  • Evaluation of the relationship between the plasma concentration of moxifloxacin and ΔΔQTc in order to demonstrate assay sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Sunu Valasseri, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Belfast, Ireland, United Kingdom